CLINICAL TRIAL: NCT06355700
Title: Hepatocellular Carcinoma Organoids to Explore Tumor Microenvironment and Test Treatment Efficacy - Hepatocellular Carcinoma Liver Organoids (HELIO)
Brief Title: Hepatocellular Carcinoma Liver Organoids
Acronym: HELIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5476
Record Dates: First submitted 2023-03-13; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hepatocellular Carcinoma (Experimental): Participants undergo to a liver biopsy, a venous blood sampling and a fecal sample collecting
  Interventions: Procedure: Liver biopsy

INTERVENTIONS:
Procedure: Liver biopsy — The liver biopsy is ultrasound-guided and target the hepatic lesions. It is performed with 18G or 19G Menghini needle. A part of bioptic sample will be used for genomic analysis. An other part of sample will be cultured to create the organoid. The organoid's cultures will be integrated with the host gut microbiota (collected by a fecal sample) and peripheral blood mononuclear cells (from venous blood sample) and they will be used for research such as molecular analysis and pharmacological tests.

SUMMARY:
The goal of this interventional study is to create hepatocellular carcinoma organoids from liver bioptic samples of individuals with hepatocellular carcinoma. The main questions it aims to answer are:

* the feasibility of hepatocellular carcinoma organoids integrated with host gut microbiota and peripheral blood mononuclear cells
* the molecular pattern of the organoid tumor microenvironment
* the in vitro therapeutic response of hepatocellular carcinoma organoids

ELIGIBILITY:
Inclusion Criteria:

* Ability to express informed consent
* Patients ≥ 18 years of age
* Radiological diagnosis of hepatocellular carcinoma (HCC)

Exclusion Criteria:

* Patients <18 years of age
* Contraindications for liver biopsy: ascites, platelet count <50.000, International Normalized Ratio (INR) >1.7
* Active viral infection
* Refusal to give informed consent for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Success rate of hepatocellular carcinoma organoids integrated with host gut microbiota and peripheral blood mononuclear cells | within 12 months
  Number of successfully created organoids from all hepatocellular carcinoma samples

SECONDARY OUTCOMES:
Analysis of hepatocellular carcinoma organoid transcriptome distribution within a reference set from The Cancer Genome Atlas | within 12 months
  Comparison between organoids transcriptome and data from The Cancer Genome Atlas
Evaluation of the concordance of somatic genetic mutations between the organoid and the original tumor | within 12 months
  DNA organoids and original tumor sample sequencing and comparison between the somatic genetic mutations found in both models
Correlation between gut microbiota community profiling and growth rate of hepatocellular carcinoma organoids | within 12 months
  Definition of microbiota composition via DNA and RNA sequencing and correlation between specific bacteria abundance and successful organoids growth
Treatment response evaluation in vitro | Day 5
  Evaluation of organoids' tumor cells survival after 5 days of chemotherapy treatment.
  Treatment will include different concentrations of sorafenib, lenvatinib, atezolizumab, bevacizumab, tremelimumab, durvalumab, regorafenib, cabozantinib. Tumor cells vitality will be assessed trough Cell TitelGlo3D Cell Viability Assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Llovet JM, Kelley RK, Villanueva A, Singal AG, Pikarsky E, Roayaie S, Lencioni R, Koike K, Zucman-Rossi J, Finn RS. Hepatocellular carcinoma. Nat Rev Dis Primers. 2021 Jan 21;7(1):6. doi: 10.1038/s41572-020-00240-3. PMID 33479224
- [Background] Huch M, Koo BK. Modeling mouse and human development using organoid cultures. Development. 2015 Sep 15;142(18):3113-25. doi: 10.1242/dev.118570. PMID 26395140
- [Background] Kretzschmar K. Cancer research using organoid technology. J Mol Med (Berl). 2021 Apr;99(4):501-515. doi: 10.1007/s00109-020-01990-z. Epub 2020 Oct 14. PMID 33057820
- [Background] Broutier L, Mastrogiovanni G, Verstegen MM, Francies HE, Gavarro LM, Bradshaw CR, Allen GE, Arnes-Benito R, Sidorova O, Gaspersz MP, Georgakopoulos N, Koo BK, Dietmann S, Davies SE, Praseedom RK, Lieshout R, IJzermans JNM, Wigmore SJ, Saeb-Parsy K, Garnett MJ, van der Laan LJ, Huch M. Human primary liver cancer-derived organoid cultures for disease modeling and drug screening. Nat Med. 2017 Dec;23(12):1424-1435. doi: 10.1038/nm.4438. Epub 2017 Nov 13. PMID 29131160
- [Background] Nuciforo S, Fofana I, Matter MS, Blumer T, Calabrese D, Boldanova T, Piscuoglio S, Wieland S, Ringnalda F, Schwank G, Terracciano LM, Ng CKY, Heim MH. Organoid Models of Human Liver Cancers Derived from Tumor Needle Biopsies. Cell Rep. 2018 Jul 31;24(5):1363-1376. doi: 10.1016/j.celrep.2018.07.001. PMID 30067989
- [Background] Ponziani FR, Bhoori S, Castelli C, Putignani L, Rivoltini L, Del Chierico F, Sanguinetti M, Morelli D, Paroni Sterbini F, Petito V, Reddel S, Calvani R, Camisaschi C, Picca A, Tuccitto A, Gasbarrini A, Pompili M, Mazzaferro V. Hepatocellular Carcinoma Is Associated With Gut Microbiota Profile and Inflammation in Nonalcoholic Fatty Liver Disease. Hepatology. 2019 Jan;69(1):107-120. doi: 10.1002/hep.30036. Epub 2018 Jul 10. PMID 29665135